CLINICAL TRIAL: NCT02131402
Title: Non-Dispensing Fitting Study Comparing the Clinical Performance of Hydrogel vs. Silicone Hydrogel Sphere Design Contact Lenses
Brief Title: Clinical Performance of Hydrogel vs. Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EX-MKTG-47
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- enfilcon A / omafilcon A (Experimental): Participants wear a pair of lenses, with a test lens in one eye and a control lens in the contra lateral eye. After approximately 1 hour of lens wear, the lenses will be removed and the next pair will be inserted. This will be repeated for a total of three pairs of lenses.
  Interventions: Device: omafilcon A
- enfilcon A / ocufilcon D (Active Comparator): Participants wear a pair of lenses, with a test lens in one eye and a control lens in the contra lateral eye. After approximately 1 hour of lens wear, the lenses will be removed and the next pair will be inserted. This will be repeated for a total of three pairs of lenses.
  Interventions: Device: ocufilcon D
- enfilcon A / methafilcon A (Active Comparator): Participants wear a pair of lenses, with a test lens in one eye and a control lens in the contra lateral eye. After approximately 1 hour of lens wear, the lenses will be removed and the next pair will be inserted. This will be repeated for a total of three pairs of lenses.
  Interventions: Device: methafilcon A

INTERVENTIONS:
Device: ocufilcon D — Contralateral pair of study lenses. Test lens (enfilcon A) in one eye and a control lens (ocufilcon D) in the contra lateral eye.
  Other Names: Hydrogel Contact Lens
  Arms: enfilcon A / ocufilcon D
Device: omafilcon A — Contralateral pair of study lenses. Test lens (enfilcon A) in one eye and a control lens (omafilcon A) in the contra lateral eye.
  Other Names: Hydrogel Contact Lens
  Arms: enfilcon A / omafilcon A
Device: methafilcon A — Contralateral pair of study lenses. Test lens (enfilcon A) in one eye and a control lens (methafilcon A) in the contra lateral eye.
  Other Names: Hydrogel Contact Lens
  Arms: enfilcon A / methafilcon A

SUMMARY:
The aim of this non-dispensing fitting study is to evaluate the subjective comfort, lens handling, lens fitting characteristics and visual acuity of different hydrogel lens designs versus silicone hydrogel lenses

DETAILED DESCRIPTION:
This is a 60-subject, double masked, randomized, contra lateral, non-dispensing fitting trial comparing different lens materials (hydrogel vs silicone hydrogel). It is anticipated that this study will involve 2 visits, for each lens pair, as follows: Visits: V1 (lens dispensing), V2 (1 hour post lens settling). Each subject will be randomized to wear the test and control lenses in a series of three short fitting comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft CL (Contact Lens) wearer
* Has a CL spherical prescription between - 1.00 and - 10.00 (inclusive)
* Has a spectacle cylinder up to 0.75D (Diopter) in each eye.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter
* Patient contact lens refraction should fit within the available parameters of the study lenses
* Is willing to comply with the wear schedule
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has never worn contact lenses before.
* Currently wears rigid gas permeable contact lenses.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has a CL prescription outside the range of - 1.00 to -10.00D
* Has a spectacle cylinder ≥1.00D of cylinder in either eye.
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities.
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montés-Mico, OD MPhil PhD, Principal Investigator — Optics Department, University of Valencia
Locations (1):
- Optometry Research Group (GIO) Optics Department, University of Valencia, Valencia, Spain

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 60 subjects enrolled and fitted with the study lenses. All sixty subjects completed the trial (i.e. no discontinuations).
Groups:
- Overall Participants Flow: Participants wear a pair of lenses, with a test lens in one eye and a control lens in the contra lateral eye. After approximately 1 hour of lens wear, the lenses will be removed and the next pair will be inserted. This will be repeated for a total of three pairs of lenses.
  omafilcon A/ocufilcon D/methafilcon A: Contralateral pair of study lenses. Test lens (enfilcon A) in one eye and a control lens (omafilcon A)/(ocufilcon D)/(methafilcon A)in the contra lateral eye.
Period: Overall Study
Arm/Group | Overall Participants Flow
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Enfilcon A / Omafilcon A/Ocufilcon D/Methafilcon A: Participants wear a pair of lenses, with a test lens in one eye and a control lens in the contra lateral eye. After approximately 1 hour of lens wear, the lenses will be removed and the next pair will be inserted. This will be repeated for a total of three pairs of lenses.
  Contralateral pair of study lenses. Test lens (enfilcon A) in one eye and a control lens (omafilcon A) in the contra lateral eye. Test lens (enfilcon A) in one eye and a control lens (ocufilcon D) in the contralateral eye. Test lens (enfilcon A) in one eye and a control lens (methafilcon A) in the contra lateral eye.
Arm/Group | Enfilcon A / Omafilcon A/Ocufilcon D/Methafilcon A
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.78 (5.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Participant's Subjective Rating for Lens Handling - Enfilcon A / Omafilcon A
Description: Surveyed after 1 hour of lens wear for each lens at lens removal Pair #1 (1 hour). Rated by questionnaires (0= Very difficult 0-100, 100= very easy).
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Participants surveyed after 1 hour of lens wear. Wearing Enfilcon A in one eye.
- Omafilcon A: Participants surveyed after 1 hour of lens wear. Wearing Omafilcon A in the contralateral eye.
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 97 (8.2) | 84 (20.2)

2. Primary Outcome: Participant's Subjective Rating for Lens Handling - Enfilcon A / Ocufilcon D
Description: Surveyed after 1 hour of lens wear for each lens at lens removal for Pair #2 (1 hour). Rated by questionnaires (0=Very difficult 0-100, 100= very easy).
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Wearing Enfilcon A in one eye. Surveyed after 1 hour of lens wear for each lens at lens removal for Pair #2.
- Ocufilcon D: Wearing Ocufilcon D in the contralateral eye. Surveyed after 1 hour of lens wear for each lens at lens removal for Pair #2
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
units on a scale | 96 (8.9) | 90 (13.7)

3. Primary Outcome: Participant's Subjective Rating for Lens Handling - Enfilcon A / Methafilcon A
Description: Surveyed after 1 hour of lens wear for each lens at lens removal Pair #3. Rated by questionnaires (0-100 0=Very difficult, 100= very easy).
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Wearing Enfilcon A in one eye. Surveyed after 1 hour of lens wear for each lens at lens removal Pair #3.
- Methafilcon A: Wearing Methafilcon A in the contralateral eye. Surveyed after 1 hour of lens wear for each lens at lens removal Pair #3.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 97 (6.5) | 86 (17.7)

4. Primary Outcome: Participants Subjective Rating for Lens Comfort - Enfilcon A / Ocufilcon D
Description: Surveyed after insertion of each lens Pair #2 (at insertion). Rated by Questionnaire (0-100,0=Can't be worn and causes pain, 100=can't feel).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Wearing Enfilcon A in one eye. Surveyed after insertion of each lens Pair #2 (at insertion).
- Ocufilcon D: Wearing Ocufilcon D in the contra lateral eye. Surveyed after insertion of each lens Pair #2 (at insertion).
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
units on a scale | 94 (9.3) | 82 (18.6)

5. Primary Outcome: Participant's Subjective Rating for Lens Comfort - Enfilcon A / Omafilcon A
Description: Surveyed after insertion of each lens at baseline visit for Pair #1. Rated by questionnaires (0-100, 0-Can't be worn and causes pain,100= can't feel).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Participants surveyed at baseline, wearing Enfilcon A in one eye
- Omafilcon A: Participants surveyed at baseline, wearing Omafilcon A in the contra lateral eye.
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 94 (8.5) | 73 (17.0)

6. Primary Outcome: Participant's Subjective Rating for Lens Comfort - Enfilcon A / Methafilcon A
Description: Surveyed after insertion Pair #3 (baseline). Rated by questionnaires (0-100, 0-Can't be worn, 100= can't feel).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Wearing Enfilcon A in one eye. Participants surveyed at insertion.
- Methafilcon A: Wearing Methafilcon A in the contra lateral eye. Participants surveyed at insertion.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 94 (9.3) | 76 (18.7)

7. Primary Outcome: Participant's Subjective Rating for Lens Comfort - Enfilcon A / Omafilcon A
Description: Surveyed after 1 hour post settling for Pair #1. Rated by questionnaires (0-100, 0= Can't be worn and causes pain, 100= can't feel).
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Participants surveyed after 1 hour post settling, wearing Enfilcon A in one eye
- Omafilcon A: Participants surveyed after 1 hour post settling, wearing Omafilcon A in contralateral eye
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 98 (4.2) | 76 (16.4)

8. Primary Outcome: Participant's Subjective Rating for Lens Comfort - Enfilcon A / Ocufilcon D
Description: Surveyed after 1 hour post settling for Pair #2. Rated by questionnaires (0-100 0=Can't be worn and causes pain, 100= can't feel).
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Wearing Enfilcon A in one eye. Surveyed after 1 hour post settling for Pair #2
- Ocufilcon D: Wearing Ocufilcon D in the contra lateral eye. Surveyed after 1 hour post settling for Pair #2.
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
units on a scale | 96 (6.1) | 83 (18.6)

9. Primary Outcome: Participant's Subjective Rating for Lens Comfort - Enfilcon A / Methafilcon A
Description: Surveyed after 1 hour post settling for Pair #3. Rated by questionnaires (0-100,0=Can't be worn and causes pain 100= can't feel).
Time Frame: 1 hours post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Methafilcon A: Participants surveyed after 1 post settling hour, wearing Methafilcon A in the contra lateral eye.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 96 (6.7) | 78 (17.7)

10. Primary Outcome: Participants Subjective Rating for Lens Comfort Preference - Enfilcon A / Omafilcon A
Description: Surveyed after insertion of each lens Pair #1 at (Baseline visit). Rated by questionnaire (4 possible ratings: Strong Enfilcon A, Slight Enfilcon A, No preference, Slight Omafilcon A, Strong Omafilcon A).
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Groups:
- Enfilcon A: Subject after insertion of Pair #1 at baseline wearing Enfilcon A in one eye
- Omafilcon A: Subject after insertion of Pair #1 at baseline wearing Omafilcon A in the contralateral eye.
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
percentage of subjects
  Strong Enfilcon A | 66.7 | 0.0
  Slight Enfilcon A | 16.7 | 0.0
  No Preference | 10.0 | 0.0
  Slight Omafilcon A | 0.0 | 6.7
  Strong Omafilcon A | 0.0 | 0.0

11. Primary Outcome: Participants Subjective Rating for Lens Comfort Preference - Enfilcon A / Ocufilcon D
Description: Surveyed at insertion of each lens Pair #2 by questionnaire (4 possible ratings: Strong Enfilcon A, Slight Enfilcon A, No preference, Slight Ocufilcon D, Strong Ocufilcon D).
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Groups:
- Enfilcon A: Wearing Enfilcon A in one eye. Surveyed at insertion of each lens Pair #2.
- Ocufilcon D: Wearing Ocufilcon D in the contralateral eye. Surveyed at insertion of each lens Pair #2.
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
percentage of subjects
  Strong Enfilcon A | 38 | 0
  Slight Enfilcon A | 22 | 0
  No Preference | 35 | 0
  Slight Ocufilcon D | 0 | 5
  Strong Ocufilcon D | 0 | 0

12. Primary Outcome: Participants Subjective Rating for Lens Comfort Preference - Enfilcon A / Methafilcon A
Description: Surveyed after insertion of each lens for Pair #3. Rated by questionnaire (4 possible ratings: Strong Enfilcon A, Slight Enfilcon A, No preference, Slight Methafilcon A, Strong Methafilcon A).
Time Frame: Baseline
Measure: Number; unit: percentage of eyes
Groups:
- Enfilcon A: Subject surveyed after insertion of each lens for Pair #3 wearing Enfilcon A in one eye
- Methafilcon A: Subject surveyed after insertion of each lens for Pair #3 wearing Methafilcon A in the contralateral eye.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
percentage of eyes
  Strong Enfilcon A | 55.0 | 0.0
  Slight Enfilcon A | 18.3 | 0.0
  No Preference | 18.3 | 0.0
  Slight Methafilcon A | 0.0 | 5.0
  Strong Methfilcon A | 0.0 | 3.3

13. Primary Outcome: Participant's Subjective Rating for Lens Comfort Preference - Enfilcon A / Omafilcon A
Description: Surveyed after 1 hour post settling (1 hour) of lens wear for Pair #1. Rated by subjects preference for test lens or control lens (Strong Enfilcon A, Slight Enfilcon A, No preference, Slight Omafilcon A, Strong Omafilcon A).
Time Frame: 1 hour post settling
Measure: Number; unit: percentage of subjects
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
percentage of subjects
  Strong Enfilcon A | 67 | 0
  Slight Enfilcon A | 20 | 0
  No preference | 13 | 0
  Slight Omafilcon A | 0 | 0
  Strong Omafilcon A | 0 | 0

14. Primary Outcome: Participant's Subjective Rating for Lens Comfort Preference - Enfilcon A / Ocufilcon D
Description: Surveyed after 1 hour post settling for Pair #2. Rated by questionnaire (4 possible ratings: Strong Enfilcon A, Slight Enfilcon A, No preference, Slight Ocufilcon D, Strong Ocufilcon D).
Time Frame: 1 hour post settling
Measure: Number; unit: percentage of subjects
Groups:
- Enfilcon A: Wearing Enfilcon A in one eye. Surveyed after 1 hour post settling.
- Ocufilcon D: Wearing Ocufilcon D in contralateral eye. Surveyed after 1 hour post settling.
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
percentage of subjects
  Strong Enfilcon A | 42 | 0
  Slight Enfilcon A | 18 | 0
  No Preference | 35 | 0
  Slight Ocufilcon D | 0 | 5
  Strong Ocufilcon D | 0 | 0

15. Primary Outcome: Participant's Subjective Rating for Lens Comfort Preference - Enfilcon A / Methafilcon A
Description: Surveyed after 1 hour post settling for Pair #3. Rated by questionnaire (4 possible ratings: Strong Enfilcon A, Slight Enfilcon A, No preference, Slight Methafilcon A, Strong Methafilcon A).
Time Frame: 1 hour post settling
Measure: Number; unit: percentage of subjects
Groups:
- Enfilcon A: Wearing Enfilcon A in one eye, surveyed at 1 hour post settling.
- Methafilcon A: Wearing Methafilcon A in the contralateral eye, surveyed at 1 hour post settling.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
percentage of subjects
  Strong Enfilcon A | 53 | 0
  Slight Enfilcon A | 22 | 0
  No Preference | 18 | 0
  Slight Methafilcon A | 0 | 7
  Strong Methafilcon A | 0 | 0

16. Primary Outcome: Eye Care Practitioner's Objective Assessment of Lens Fit, Post-blink Movement, and Primary Gaze Lag - Enfilcon A / Omafilcon A
Description: Assessed after 1 hour post settling of lens wear for Pair #1. Slit lamp (0-4, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement)
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Assessed after 1 hour post settling. Post-blink movement, wearing Enfilcon A in one eye.
- Omafilcon A: Assessed after 1 hour post settling. Post-blink movement, wearing Omafilcon A in contralateral eye.
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 2.0 (0) | 2.0 (0)

17. Primary Outcome: Eye Care Practitioner's Objective Assessment of Lens Fit, Post-blink Movement, and Primary Gaze Lag - Enfilcon A / Ocufilcon D
Description: Assessed after 1 hour post settling for Pair #2. (0-4, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement)
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ocufilcon D: Assessed after 1 hour post settling. Post-blink movement, wearing Ocufilcon D in contralateral eye.
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
units on a scale | 2.0 (0) | 2.0 (0)

18. Primary Outcome: Eye Care Practitioner's Objective Assessment of Lens Fit, Post-blink Movement, and Primary Gaze Lag - Enfilcon A / Methafilcon A
Description: Assessed after 1 hour post settling for Pair #3. (0-4, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement)
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Assessed at 1 hour post settling. Post-blink movement, wearing Enfilcon A in one eye.
- Methafilcon A: Assessed at 1 hour post settling. Post-blink movement, wearing Ocufilcon D in contralateral eye.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 2.0 (0) | 2.0 (0)

19. Primary Outcome: Eye Care Practitioner's Objective Assessment of Lens Fit, Tightness Push-up Test - Enfilcon A / Omafilcon A
Description: Assessed after 1 hour post settling of lens wear for Pair #1. Slit lamp. (0%-100%, continuous scale where 100%=no movement, 50%=optimum, 0%=Falls from cornea without lid support).
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Assessed after 1 hour post settling. Push up test, wearing Enfilcon A in one eye.
- Omafilcon A: Assessed after 1 hour post settling. Push up test, wearing Omafilcon A in contralateral eye.
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 50 (1.8) | 50 (1.8)

20. Primary Outcome: Eye Care Practitioner's Objective Assessment of Lens Fit, Tightness Push-up Test - Enfilcon A / Ocufilcon D
Description: Assessed after 1 hour post settling for Pair #2, (0%-100%, continuous scale where 100%=no movement, 50%=optimum, 0%=Falls from cornea without lid support).
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ocufilcon D: Assessed after 1 hour post settling. Push up test, wearing Ocufilcon D in contralateral eye.
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
units on a scale | 50 (0.65) | 50 (0.65)

21. Primary Outcome: Eye Care Practitioner's Objective Assessment of Lens Fit, Tightness Push-up Test - Enfilcon A / Methafilcon A
Description: Assessed after 1 hour post settling for Pair #3. (Scale 0%-100%, 0%-100%, continuous scale where 100%=no movement, 50%=optimum, 0%=Falls from cornea without lid support)
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Assessed at 1 hour post settling. Push up test, wearing Enfilcon A in one eye.
- Methafilcon A: Assessed at 1 hour post settling. Push up test, wearing Methafilcon A in contralateral eye.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 50 (0.91) | 50 (0.65)

22. Primary Outcome: Eye Care Practitioner's Objective Assessment of Lens Fit, Centration - Enfilcon A / Omafilcon A
Description: Assessed after 1 hour post settling of lens wear for Pair #1. (4 possible ratings: optimum, Decentration acceptable, Decentration unacceptable).
Time Frame: 1 hour post settling
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Enfilcon A: Assessed after 1 hour post settling wearing Enfilcon A in one eye.
- Omafilcon A: Assessed after 1 hour post settling, wearing Omafilcon A in contralateral eye
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Optimum | 100 | 100
  Decentration acceptable | 0 | 0
  Decentration unacceptable | 0 | 0

23. Primary Outcome: Eye Care Practitioner's Objective Assessment of Lens Fit, Centration - Enfilcon A / Ocufilcon D
Description: Assessed after 1 hour post settling for Pair #2. (4 possible ratings: optimum, Decentration acceptable, Decentration unacceptable)
Time Frame: 1 hour post settling
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Enfilcon A: Assessed after 1 hour post settling, wearing Enfilcon A in one eye.
- Ocufilcon D: Assessed after 1 hour post settling, wearing Ocufilcon D in contralateral eye.
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Optimum | 100 | 100
  Decentration Acceptable | 0 | 0
  Decentration Unacceptable | 0 | 0

24. Primary Outcome: Eye Care Practitioner's Objective Assessment of Lens Fit, Centration - Enfilcon A / Methafilcon A
Description: Assessed after 1 hour post settling for Pair #3, (4 possible ratings: optimum, Decentration acceptable, Decentration unacceptable)
Time Frame: 1 hour post settling
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Enfilcon A: Assessed at 1 hour post settling, wearing Enfilcon A in one eye.
- Methafilcon A: Assessed at 1 hour post settling, wearing Methafilcon A in contralateral eye.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Optimum | 100 | 100
  Decentration acceptable | 0 | 0
  Decentration unacceptable | 0 | 0

25. Primary Outcome: Participant's Subjective Rating for Stinging/Burning - Enfilcon A / Omafilcon A
Description: Surveyed after insertion of each lens for Pair #1 at baseline visit. Rated by questionnaires (0-100, 0=no sensation of stinging/burning, 100= extreme stinging).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Omafilcon A: Participants surveyed at baseline, wearing Omafilcon A in contralateral eye
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 2.6 (6.00) | 18 (22.6)

26. Primary Outcome: Participant Subjective Rating for Stinging/Burning - Enfilcon A / Ocufilcon D
Description: Surveyed after insertion of each lens Pair #2 at baseline. Rated by questionnaires (0-100,0=no sensation of stinging/burning 100=extreme stinging)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Surveyed after insertion at baseline, wearing Enfilcon A in one eye.
- Ocufilcon D: Surveyed after insertion at baseline, wearing Ocufilcon D in contralateral eye.
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
units on a scale | 3.3 (9.5) | 11 (20.3)

27. Primary Outcome: Participant Subjective Rating for Stinging/Burning - Enfilcon A / Methafilcon A
Description: Surveyed after insertion of each lens for Pair #3. Rated by questionnaires (0-100,0=no sensation of stinging/burning, 100=extreme stinging).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Methafilcon A: Participants surveyed at baseline, wearing Methafilcon A in contralateral eye.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 2.0 (4.0) | 15 (19.8)

28. Primary Outcome: Participants Subjective Rating for Stinging/Burning - Enfilcon A / Omafilcon A
Description: Surveyed after 1 hour of lens wear for each lens at lens removal Pair #1. Rated by questionnaires (0-100,0=no sensation of stinging/burning 100=extreme stinging).
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Participants surveyed after 1 hour wearing Enfilcon A in one eye.
- Omafilcon A: Participants surveyed after1 hour wearing Omafilcon A in contralateral eye.
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 0.6 (2.3) | 8.8 (13.4)

29. Primary Outcome: Participant's Subjective Rating for Stinging/Burning - Enfilcon A / Ocufilcon D
Description: Surveyed after 1 hour post settling for Pair #2. Rated by questionnaires (0-100,0= no sensation of stinging/burning, 100= extreme stinging).
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enfilcon A: Participants surveyed at 1 hour post settling, wearing Enfilcon A in one eye.
- Ocufilcon D: Participants surveyed at 1 hour post settling, wearing Ocufilcon D in contralateral eye.
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
units on a scale | 1.4 (3.5) | 8.8 (13.9)

30. Primary Outcome: Participant's Subjective Rating for Stinging/Burning - Enfilcon A / Methafilcon A
Description: Surveyed after 1 hour post settling for Pair #3. Rated by questionnaires (0-100,0= no sensation of stinging/burning,100= extreme stinging).
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Methafilcon A: Participants surveyed at 1 hour post settling, wearing Methafilcon A in contralateral eye.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 1.2 (3.2) | 13 (18.7)

31. Primary Outcome: Eye Care Practitioner's Objective Assessment of Binocular High Contrast Distance Visual Acuity - Enfilcon A / Omafilcon A
Description: Visual acuity assessed after insertion of each study lens, prior to dispensing contralateral pairs Pair #1. LogMAR Visual Acuity (VA) to nearest letter)
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Enfilcon A: Participants vision tested both eyes wearing enfilcon A, prior to dispensing contralateral pairs.
- Omafilcon A: Participants vision tested both eyes wearing omafilcon A, prior to dispensing contralateral pairs.
Arm/Group | Enfilcon A | Omafilcon A
Number analyzed (Participants) | 60 | 60
LogMAR | -0.041 (0.049) | -0.035 (0.055)

32. Primary Outcome: Eye Care Practitioner's Objective Assessment of Binocular High Contrast Distance Visual Acuity - Enfilcon A / Ocufilcon D
Description: Visual acuity assessed after insertion of each study lens, prior to dispensing contralateral pairs- Pair #2. LogMAR Visual Acuity (VA) to nearest letter)
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Ocufilcon D: Participants vision tested both eyes wearing ocufilcon D, prior to dispensing contralateral pairs.
Arm/Group | Enfilcon A | Ocufilcon D
Number analyzed (Participants) | 60 | 60
LogMAR | -0.041 (0.049) | -0.040 (0.049)

33. Primary Outcome: Eye Care Practitioner's Objective Assessment of Binocular High Contrast Distance Visual Acuity - Enfilcon A / Methafilcon A
Description: Visual acuity assessed after insertion of each study lens, prior to dispensing contralateral pairs- Pair #3. LogMAR Visual Acuity (VA) to nearest letter)
Time Frame: 1 hour post settling
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Methafilcon A: Participants vision tested both eyes wearing Methafilcon A, prior to dispensing contralateral pairs.
Arm/Group | Enfilcon A | Methafilcon A
Number analyzed (Participants) | 60 | 60
LogMAR | -0.041 (0.049) | -0.043 (0.050)

ADVERSE EVENTS:
Arm/Group | Enfilcon A / Omafilcon A | Enfilcon A / Ocufilcon D | Enfilcon A / Methafilcon A
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.